CLINICAL TRIAL: NCT04775615
Title: A Study on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multi-dose DDO-3055 Tablets in Healthy Subjects-Randomized, Double-blind, Dose Escalation, Placebo Controlled Phase I Clinical Trial.
Brief Title: Multi-dose, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DDO-3055 Tablets in Healthy Subjects.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DDO-3055-105
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Renal Anemia

STUDY DESIGN:
Intervention Model Description: Multi-dose, dose escalation study in healthy subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental)
  Interventions: Drug: DDO-3055 tablets；Placebo
- Treatment group B (Experimental)
  Interventions: Drug: DDO-3055 tablets；Placebo
- Treatment group C (Experimental)
  Interventions: Drug: DDO-3055 tablets；Placebo

INTERVENTIONS:
Drug: DDO-3055 tablets；Placebo — Low dose：DDO-3055 tablets for 7 days or Placebo for 7 days
  Arms: Treatment group A
Drug: DDO-3055 tablets；Placebo — Medium dose：DDO-3055 tablets for 7 days or Placebo for 7 days
  Arms: Treatment group B
Drug: DDO-3055 tablets；Placebo — High dose：DDO-3055 tablets for 7 days or Placebo for 7 days
  Arms: Treatment group C

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multi-dose DDO-3055 tablets in healthy subjects for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 18-45 years;
2. Male weight≥50kg, female weight≥45kg, and 19kg/m2≤BMI≤26kg/m2;
3. Signed informed consent.

Exclusion Criteria:

1. Allergic constitution, suspected to be allergic to the study drug or any component in the study drug;
2. A value at screening is greater than the upper limit of reference range for the following clinical laboratory parameters: AST, ALT, Total bilirubin, direct bilirubin, indirect bilirubin ；
3. Subjects with a value at screening is greater than the upper limit of reference range for serum creatinine;
4. Subjects with a positive value of HBsAg、HCV-Ab、HIV-Ab、TPPA at screening；
5. Subjects with blood loss ≥400mL within 3 months before screening;
6. Subjects has participated in a clinical trial and has received an investigational product within 3 months prior to the first dosing day in the current study.
7. Participants who are unwilling to take contraception or male subjects who cannot guarantee not to donate sperm during the trial and within 30 days after the last dose; female subjects with fertility who did not use contraception for at least 14 days before dosing;
8. Patients who had a positive blood pregnancy test and were breastfeeding at the time of screening.
9. Smokers (average daily smoking 5 or more); Subjects who consumed more than 15 grams of alcohol per day within one week prior to the screening;
10. Drug abusers or drug urine screening positive;
11. The researchers judged that the subjects had medical conditions that affected the absorption, distribution, metabolism and excretion of drugs or reduced compliance.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-03-17 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events (AE) | up to 14 days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) on Day 1 and Day 7 | Pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Peak plasma concentration (Cmax) on Day 1 and Day 7 | Pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Time to maximum plasma concentration (Tmax) on Day 1 and Day 7 | Pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post-dose
Change of endogenous erythropoietin from baseline :Day 1 and Day 7 | 0, 24 hours post dose
Change of VEGF from baseline :Day 1 and Day 7 | 0, 24 hours post dose
Change of Hb from baseline | Day1, Day7, Day14
Change of Ret from baseline | Day1, Day7, Day14
Change of Hepcidin from baseline | Day1, Day 9
Change of Ferritin from baseline | Day1, Day 9
Change of Serum Iron from baseline | Day1, Day 9